CLINICAL TRIAL: NCT03947229
Title: A Randomized Comparison of CLOpidogrel Monotherapy Versus Extended Dual-antiplatelet Therapy Beyond 12 Months After Implantation of Drug-eluting StEnts in High-risk Lesions or Patients; A-CLOSE Trial
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2019-0234
Record Dates: First submitted 2019-05-08; First posted 2019-05-13 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Coronary Artery Disease; DES
Keywords: Patients who underwent percutaneous coronary intervention with DES implantation carrying high risks for the recurrent major adverse events.; anti platelet therapy; bleeding
MeSH Terms: conditions — Coronary Artery Disease; Hemorrhage

STUDY DESIGN:
Intervention Model Description: Patients will be assigned to continue DAPT (aspirin plus clopidogrel) or to change to single antiplatelet therapy with clopidogrel (clopidogrel-alone) for further 24 months.
Masking Description: Antiplatelet drugs will be open-label and prescribed by attending physician.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clopidogrel mono-therapy (Active Comparator): After randomization, patients will receive clopidogrel monotherapy after DES implantation for 24 months.
  Interventions: Drug: Clopidogrel mono-therapy
- Dual-antiplatelet therapy (Active Comparator): Patients will receive dual antiplatelet consisting of aspirin and clopidogrel.
  Interventions: Drug: Dual-antiplatelet therapy

INTERVENTIONS:
Drug: Clopidogrel mono-therapy — Patients will receive clopidogrel (75 mg once daily) monotherapy without co-administration of aspirin for 24 months after randomization.
  Arms: Clopidogrel mono-therapy
Drug: Dual-antiplatelet therapy — Patients will receive co-administration of aspirin (100 mg/day) and clopidogrel (75 mg/day) for 24 months after randomization.
  Arms: Dual-antiplatelet therapy

SUMMARY:
We hypothesized that clopidogrel mono-therapy will not be inferior to the extended DAPT in terms of the occurrence of both ischemic and bleeding events, for lesions or patients at high risk for either ischemic or bleeding complications 12 months after drug-eluting stent (DES) implantation.

DETAILED DESCRIPTION:
Patients at high risk for either ischemic or bleeding complications, but who were stable without clinical evetns for 12 months after DES implantation will be included in this study. Eligible patients will be randomized to continue DAPT (aspirin plus clopidogrel) for further 24 months or to change to single antiplatelet therapy with clopidogrel (clopidogrel-alone). Randomization will be stratified according to 1) clinical presentation (acute coronary syndrome or stable coronary artery disease) and 2) age (≥75 or <75). Baseline clinical and angiographic characteristics, laboratory findings will be assessed at the time of randomization. All patients will provide informed consent on their own initiative. All of study subjects will be have an outpatient visit as scheduled in outpatient clinic. Occurrence of study endpoints will be documented at clinical visit or telephone interview every 6 months up to 24 months after randomization. Antiplatelet drugs will be open-label and prescribed by attending physician.

ELIGIBILITY:
Inclusion criteria (must all met)

1. Patients >19 years old
2. Patients who underwent DES implantation 12 months (-1 to +5 months) previously.
3. High risk characteristics (clinical or lesion) for ischemic events (must at least one)

High risk patients; clinical criteria

1. Acute coronary syndrome
2. Previous history of cerebrovascular accidents
3. History of peripheral artery intervention
4. Heart failure (left ventricular ejection fraction ≤40%)
5. Diabetes treated with medication
6. Chronic renal insufficiency including end-stage renal diseases

High risk lesions; angiographic or procedural criteria

1. Left main diseases
2. Bifurcation lesions
3. Chronic total occlusion
4. In-stent restenotic lesions
5. Graft lesions
6. Diffuse long lesions requiring total stent length ≥28 mm
7. Calcified lesions requiring atherectomy
8. Multivessel coronary artery disease with multiple stents
9. Small vessel disease requiring stent diameter of ≤2.5 mm

Exclusion criteria

1. Age> 80 years
2. Pregnant women or women with potential childbearing
3. Life expectancy < 1 year
4. Refusal or inability to understand of informed consent
5. Need for chronic oral anticoagulation
6. History of major bleeding within 3 months prior to randomization

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3200 (Actual)
Dates: Start 2019-08-14 (Actual); Primary Completion 2025-08-16 (Estimated); Study Completion 2026-08-16 (Estimated)

PRIMARY OUTCOMES:
Net Adverse Clinical Events (NACE) | 24 months
  The composite of all-cause of death, myocardial infarction (MI), stent thrombosis, stroke, or bleeding (BARC type 2, 3, or 5)

SECONDARY OUTCOMES:
Each component of net adverse clinical events | 24 months
All-cause or cardiovascular mortality | 24 months
Major or minor bleeding | 24 months
  Major or minor bleeding would be defined by BARC and TIMI criteria
Major adverse cardiac event | 24 months
  Major Adverse Cardiac events includes all-cause of death, myocardial infarction, stent thrombosis, or ischemia-driven target vessel revascularization
Major adverse cardiac and cerebrovascular event | 24 months
  Major adverse cardiac and cerebrovascular event includes all-cause death, myocardial infarction, stent thrombosis, stroke, or ischemia-driven target vessel revascularization

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Cardiology, Severance Cardiovascular Hospital Yonsei University College of Medicine, 250 Seongsanno, Seodaemun-gu 120-752 Seoul, South Korea, Seoul, South Korea